CLINICAL TRIAL: NCT00533819
Title: A Phase II Non Randomized Community Intervention Trial in 4 Public Sectors Schools in Karachi. Exercise Intervention in Female School Children: Effect on Blood Pressure, BMI, and Maths Scores
Brief Title: Exercise Intervention in Female School Children: Effect on Blood Pressure, Body Mass Index (BMI), and Maths Scores
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07GS006CHS; 743-CHS/ERC-07
Record Dates: First submitted 2007-09-20; First posted 2007-09-21 (Estimated); Last update posted 2008-10-15 (Estimated); Status verified 2008-10

CONDITIONS: Hypertension
Keywords: Exercise intervention; Maths Scores; Blood pressure; Female school children; Body mass index
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Other: 6 months of healthy physical activity
- 2 (No Intervention): would have routine physical activity

INTERVENTIONS:
Other: 6 months of healthy physical activity — half an hour of healthy physical activity including 20 minutes aerobic, 5 minutes warm up and cool down, 4 days a week
  Arms: 1

SUMMARY:
Healthy physical activity decreases blood pressure in young female school children. It also has effects on BMI and maths scores.

DETAILED DESCRIPTION:
* Primary Objective: To compare the effect of 6 months healthy physical activity on blood pressure in female school children (9-13 yrs) with those who have routine physical activity
* Secondary objective: To compare the effect of 6 months of healthy physical activity on body mass index and maths scores with those who have routine physical activity
* Study Design: It would be a non-randomized experimental study (community intervention trial). It is designed to test the effectiveness of exercise on reducing blood pressure and the effect on BMI and maths scores
* Setting: The study would be conducted in 4 public sector schools in Karachi.
* Study Population: The study population would be selected from 4 local public sector schools near our hospital, The Aga Khan University Hospital. Two schools would have intervention and 2 schools would serve as controls. Both groups would have a base line screening for the outcome variables and then at 6 months
* Intervention: The intervention is 30 minutes of healthy physical activity; 4-times/week would be carried out for a period of 6 months. This would be carried out by certified physical trainers who are experts in training children in aerobic exercise. Intervention group will have half an hour session on exercise motivation and its benefits. The routine activity group will have a similar session at baseline.
* Sampling technique: convenience sampling
* Sample Size : A sample size of 126 (63 in each arm) achieves 80% power to detect a difference of 4.3 mm in systolic blood pressure between the null hypothesis mean of 110.3 and an alternative hypothesis mean of 105.7 with an estimated standard deviation of 9.7 and with significance level (alpha) of 0.05 using one sided one sample t test. Assuming that there could be a 10% dropout rate we plan to take a total sample size of 140 students. We multiplied the total sample size by 2 to account for the design effect between clusters (schools) and achieved a total sample size of 280 that is 140 in each arm.
* Dependent variables or outcome variables: Primary outcome measure would be the blood pressure. Secondary outcome measures would be body composition including weight, BMI, central obesity, and maths score. Independent variable would be demographics (age, school class) and the intervention of healthy physical activity and measurement of food intake frequency

ELIGIBILITY:
Inclusion Criteria:

* Female children of age 9-11 yrs who are enrolled in the public sector school with a compound facility would be included in the study. Intervention would be offered to those only who will have normal age specific weight in percentiles.

Exclusion Criteria:

* Those who are suffering from any chronic illness due to they which cannot participate and those who are mentally or physically disabled will be excluded from the study.

Ages: 9 Years to 11 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Estimated)
Dates: Start 2007-09; Study Completion 2008-05 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | 6 months

SECONDARY OUTCOMES:
Body mass index | 6 months
Maths scores | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Aysha Almas, MBBS, FCPS, Principal Investigator — Student
Locations (1):
- 4 Public Sector Schools, Karachi, Sindh, Pakistan

REFERENCES:
- [Background] Yin Z, Gutin B, Johnson MH, Hanes J Jr, Moore JB, Cavnar M, Thornburg J, Moore D, Barbeau P. An environmental approach to obesity prevention in children: Medical College of Georgia FitKid Project year 1 results. Obes Res. 2005 Dec;13(12):2153-61. doi: 10.1038/oby.2005.267. PMID 16421350
- [Derived] Almas A, Islam M, Jafar TH. School-based physical activity programme in preadolescent girls (9-11 years): a feasibility trial in Karachi, Pakistan. Arch Dis Child. 2013 Jul;98(7):515-9. doi: 10.1136/archdischild-2012-303242. Epub 2013 May 9. PMID 23661575